CLINICAL TRIAL: NCT06627049
Title: Virtual Reality Implantation in Paediatric Rehabilitation (IMPLANT-VR4 CHILD)
Acronym: IMPLANT-VR4
Status: Recruiting | Type: Observational
Sponsor: Fondation Ildys (Other)
Responsible Party: Sponsor
Other Study IDs: RI2024_008
Record Dates: First submitted 2024-09-23; First posted 2024-10-04 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Children with Undergoing Rehabilitation
Keywords: Virtual Reality; Active Video Games; Paediatric rehabilitation; Implementation Science; Action Research
MeSH Terms: interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Rehabilitation professionals: Pediatric rehabilitation professionals
  Interventions: Other: Focus group; Other: Implementing facilitating strategies
- Decision makers: healthcare managers or directors
  Interventions: Other: Interviews
- Children: Children in paediatric rehabilitation services
  Interventions: Other: Focus group; Other: Implementing facilitating strategies

INTERVENTIONS:
Other: Focus group — Focus group to evaluate the facilitators and barriers to the use of virtual reality.
  Groups: Children; Rehabilitation professionals
Other: Implementing facilitating strategies — Implement strategies to facilitate the integration of virtual reality into rehabilitation sessions.
  Groups: Children; Rehabilitation professionals
Other: Focus group — Evaluate the strategies used to facilitate VR implementation.
  Groups: Children; Rehabilitation professionals
Other: Interviews — Interviews to evaluate the facilitators and barriers to the use of virtual reality.
  Groups: Decision makers
Other: Interviews — Evaluate the strategies used to facilitate VR implementation.
  Groups: Decision makers

SUMMARY:
Virtual Reality Implementation in Paediatric Rehabilitation (IMPLANT-VR 4 CHILD) Virtual Reality (VR) and Active Video Games (AVG) are promising devices for children in need of rehabilitation. VR and AVG have been widely studied in research, with promising results in a number of areas, including motor function, cognitive function, pain management and attention disorders.

However, despite these promising results and the enthusiasm they generate in research, VR and AVG are rarely used in clinical practice, particularly in the paediatric services of Ty Yann and Perharidy of the ILDYS Foundation. There is a strong demand from professionals for these tools to be better integrate these devices into their clinical practice.

The project is to conduct an action research with rehabilitation professionals, health managers and children in need of rehabilitation in order to facilitate the implementation of VR and AVG in the paediatric rehabilitation services of Ty Yann and Perharidy. Firstly, the facilitators and barriers present in these services will be identified. Then, specific strategies to facilitate the implementation of VR will be used. Finally, the impact of these strategies on the use of VR will be evaluated.

DETAILED DESCRIPTION:
Children with chronic conditions and rehabilitation needs may require long periods of care. Some rehabilitation interventions can cause stress, anxiety or pain and may be unmotivating for children. However, in the context of motor learning, for example, current scientific research supports the intensification of training.

Motivation is a fundamental part of rehabilitation treatment. Sometimes the length of treatment can lead to a lack of motivation. If motivation decreases in children, this may lead to a reduction in the intensity required to be effective in rehabilitation. Finding efficient solutions to facilitate the rehabilitation process is therefore a major challenge. Virtual reality (VR) may be interesting to increase the duration of motor rehabilitation while maintaining motivation.

VR is a promising tool to address these challenges. VR can be defined as the digital simulation of a virtual environment with which the user can interact using our own movements. Immersive VR devices use a head-mounted display that allows full visual immersion in the virtual environment. Non-immersive VR devices involve two-dimensional virtual environment in flat-screen displays, and include the category of AVG. It has been studied in many areas of paediatric rehabilitation (motor function, pain management, attention disorders, cognitive function). For example, in motor rehabilitation, the playful aspect of VR helps to maintain children's motivation, while facilitating motor learning. VR games can be played at high intensity. Rehabilitation goals can also be set by the child when using VR, increasing the effectiveness of rehabilitation management.

The aim of implementation science is to facilitate the integration and use of evidence in clinical practice. There are often differences between research findings and the methods used in clinical practice. It often takes several years for research findings to be implemented in clinical practice. It is estimated that it takes about 17 years in some fields for a scientific discovery to be used in clinical practice. There are a number of factors that may explain this long delay. First of all, there are several stages in the research process to develop practice guidelines. These stages are relatively long. In addition, clinicians often have little time to read newly published data, and these data are not always easily accessible.

VR is still rarely used into routine clinical practice, despite promising results and the enthusiasm it generates in research. There are barriers, such as the time required to prepare sessions and a lack of knowledge about the devices. Some barriers to the implementation of VR are common to several rehabilitation centres, and are frequently found in the literature, while others are specific to one rehabilitation centre. In order to address the specific barriers, it is necessary to identify them within the rehabilitation centre itself.

Several studies have identified the facilitators and barriers present among rehabilitation professionals. To our knowledge, this work has not been carried out among decision makers (managers and directors of rehabilitation centres), nor among children undergoing rehabilitation. However, the facilitators and barriers to the implementation of VR may come from different levels within the rehabilitation centre. For example, national care policies, funding for VR, the organisation of services, and the beliefs of professionals and children are all factors that can influence the way care is provided and whether or not VR devices are used. Therefore, in order to be as effective and comprehensive as possible when implementing VR in paediatric rehabilitation, it is recommended to consider the facilitators and barriers related to rehabilitation professionals, decision makers and children.

The ILDYS Foundation is a rehabilitation centre. Every week, this institution welcomes around 200 children with disabilities in its different services, located in two sites, Perharidy and Ty Yann. Both sites provide rehabilitation for children and adolescents with chronic conditions that limit their activities and participation and therefore require rehabilitation treatment.

There is a demand from rehabilitation professionals and the decision makers to facilitate the integration of VR, which is currently little used in the services. However, during informal discussions, many barriers were mentioned that could explain the lack of use of VR during rehabilitation sessions.

Action research can be defined as work carried out in collaboration between researchers and participants. This collaboration makes it possible to involve clinicians, decision makers and patients in the study, which can facilitate the implementation of new care strategies.

The main objective of this project is to improve the use of VR in the Ty Yann and Perharidy paediatric rehabilitation centre. In order to carry out this implementation project, the study is divided into three stages:

* First, the facilitators and barriers that exist in the services at Ty Yann and Perharidy will be identified. Several focus groups with rehabilitation professionals, and children in rehabilitation in Ty Yann and Perharidy will be conducted. The investigator will conduct some interviews with decision makers at the ILDYS Foundation. The investigator will collect socio-demographic data from the participants in order to characterise the population involved in this research project. The investigator will also collect data on the use of VR and the ease of use of VR by rehabilitation professionals. Tne investigator will collect socio-demographic data from the participants in order to characterise the population taking part in this research project. Data will also be collected on the use of VR and the ease of use of VR by rehabilitation professionals.
* Secondly, specific strategies to improve the use of VR according to the focus group and interview responses will be implemented.
* Thirdly, the strategies in terms of the number of uses of the VR devices will be evaluated. On the other hand, focus groups and interviews will be used to collect the views of rehabilitation professionals, decision makers and children on the implemented strategies.

ELIGIBILITY:
Inclusion Criteria for rehabilitation professionals::

* Rehabilitation professional
* Be fluent in French.
* Work in the paediatric wards at Ty Yann or Perharidy.
* Consent to data processing

Inclusion Criteria for Children :

* Be aged between 6 and 18.
* Be fluent in French.
* Have received rehabilitation treatment in the Ty Yann or Perharidy paediatric services.
* Have already used virtual reality in a rehabilitation session.
* Have the consent of the child and his/her legal representative to take part in the study.

Inclusion Criteria for decision makers:

* Work at the ILDYS Foundation as a health executive or within the management team.
* Be fluent in French.
* Consent to data processing

Exclusion Criteria:

* Not being able to understand focus group or interview questions.
* Not being able to communicate during focus groups or interviews.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric rehabilitation professionals ; Children in paediatric rehabilitation services ; Decision makers of the rehabilitation centre
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Form of the number of uses per week | October 2024 - november 2025
  This form will be used to record the use of VR tools in paediatric rehabilitation, in order to extract the number of times VR devices are used per week. Thanks to this form, we will be able to know if the use of VR devices has increased after the implementation of the strategies. This form will be introduced before, during and after the implementation of the strategies in order to quantify changes in the use of VR. The professionals will complete this form at each session.
Focus group and interviews based on the Consolidated Framework for Implementation Research (CFIR) | October 2024 - november 2025
  The CFIR is a conceptual framework used to guide the implementation process. We will use focus groups and interviews to assess facilitators and barriers to the use and the implementation of VR. These results will help us to implement specific strategies. Focus group and interviews will be used to evaluate the strategies. Qualitative methods will be used in Stage 1 to select the strategies to be implemented to improve the use of VR. In Stage 3, the focus group and interviews will be used to gather the views of professionals, decision makers and children on the strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Jéromine HERVO, Principal Investigator — Fondation Ildys
Locations (2):
- France (2):
  - Fondation ILDYS, Site de Ty Yann, Brest
  - Fondation ILDYS, Site de Perharidy, Roscoff

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordeiro L, Soares CB. Action research in the healthcare field: a scoping review. JBI Database System Rev Implement Rep. 2018 Apr;16(4):1003-1047. doi: 10.11124/JBISRIR-2016-003200. PMID 29634517
- [Background] Waltz TJ, Powell BJ, Fernandez ME, Abadie B, Damschroder LJ. Choosing implementation strategies to address contextual barriers: diversity in recommendations and future directions. Implement Sci. 2019 Apr 29;14(1):42. doi: 10.1186/s13012-019-0892-4. PMID 31036028
- [Background] Glegg SMN, Holsti L, Stanton S, Hanna S, Velikonja D, Ansley B, Sartor D, Brum C. Evaluating change in virtual reality adoption for brain injury rehabilitation following knowledge translation. Disabil Rehabil Assist Technol. 2017 Apr;12(3):217-226. doi: 10.3109/17483107.2015.1111944. Epub 2016 Jan 10. PMID 28508725
- [Background] Levac D, Glegg SM, Sveistrup H, Colquhoun H, Miller PA, Finestone H, DePaul V, Harris JE, Velikonja D. A knowledge translation intervention to enhance clinical application of a virtual reality system in stroke rehabilitation. BMC Health Serv Res. 2016 Oct 6;16(1):557. doi: 10.1186/s12913-016-1807-6. PMID 27716179
- [Background] Kouijzer MMTE, Kip H, Bouman YHA, Kelders SM. Implementation of virtual reality in healthcare: a scoping review on the implementation process of virtual reality in various healthcare settings. Implement Sci Commun. 2023 Jun 16;4(1):67. doi: 10.1186/s43058-023-00442-2. PMID 37328858
- [Background] Banerjee-Guenette P, Bigford S, Glegg SMN. Facilitating the Implementation of Virtual Reality-Based Therapies in Pediatric Rehabilitation. Phys Occup Ther Pediatr. 2020;40(2):201-216. doi: 10.1080/01942638.2019.1650867. Epub 2019 Aug 16. PMID 31416381
- [Background] Levac D, Glegg S, Colquhoun H, Miller P, Noubary F. Virtual Reality and Active Videogame-Based Practice, Learning Needs, and Preferences: A Cross-Canada Survey of Physical Therapists and Occupational Therapists. Games Health J. 2017 Aug;6(4):217-228. doi: 10.1089/g4h.2016.0089. PMID 28816511
- [Background] Green LW, Ottoson JM, Garcia C, Hiatt RA. Diffusion theory and knowledge dissemination, utilization, and integration in public health. Annu Rev Public Health. 2009;30:151-74. doi: 10.1146/annurev.publhealth.031308.100049. PMID 19705558
- [Background] Glasziou P, Haynes B. The paths from research to improved health outcomes. Evid Based Nurs. 2005 Apr;8(2):36-8. doi: 10.1136/ebn.8.2.36. No abstract available. PMID 15830412
- [Background] Olswang LB, Prelock PA. Bridging the Gap Between Research and Practice: Implementation Science. J Speech Lang Hear Res. 2015 Dec;58(6):S1818-26. doi: 10.1044/2015_JSLHR-L-14-0305. PMID 26262822
- [Background] Kanitkar A, Parmar ST, Szturm TJ, Restall G, Rempel GR, Sepehri N, Naik N. Evaluation of a computer game-assisted rehabilitation program for manual dexterity of children with cerebral palsy: Feasibility randomized control trial. PM R. 2023 Oct;15(10):1280-1291. doi: 10.1002/pmrj.12947. Epub 2023 Jun 28. PMID 36655404
- [Background] Gehringer JE, Fortin E, Surkar SM, Hao J, Pleiss M, Jensen-Willett S. Hand-Arm Bimanual Intensive Training in Virtual Reality: A Feasibility Study. Pediatr Phys Ther. 2023 Jan 1;35(1):85-91. doi: 10.1097/PEP.0000000000000975. Epub 2022 Dec 2. PMID 36459077
- [Background] Reifenberg G, Gabrosek G, Tanner K, Harpster K, Proffitt R, Persch A. Feasibility of Pediatric Game-Based Neurorehabilitation Using Telehealth Technologies: A Case Report. Am J Occup Ther. 2017 May/Jun;71(3):7103190040p1-7103190040p8. doi: 10.5014/ajot.2017.024976. PMID 28422630
- [Background] Tatla SK, Sauve K, Virji-Babul N, Holsti L, Butler C, Van Der Loos HF. Evidence for outcomes of motivational rehabilitation interventions for children and adolescents with cerebral palsy: an American Academy for Cerebral Palsy and Developmental Medicine systematic review. Dev Med Child Neurol. 2013 Jul;55(7):593-601. doi: 10.1111/dmcn.12147. Epub 2013 Mar 29. PMID 23550896
- [Background] Monge Pereira E, Molina Rueda F, Alguacil Diego IM, Cano de la Cuerda R, de Mauro A, Miangolarra Page JC; CONSOLIDER-Ingenio 2010. Use of virtual reality systems as proprioception method in cerebral palsy: clinical practice guideline. Neurologia. 2014 Nov-Dec;29(9):550-9. doi: 10.1016/j.nrl.2011.12.004. Epub 2012 Feb 17. English, Spanish. PMID 22341675
- [Background] Warnier N, Lambregts S, Port IV. Effect of Virtual Reality Therapy on Balance and Walking in Children with Cerebral Palsy: A Systematic Review. Dev Neurorehabil. 2020 Nov;23(8):502-518. doi: 10.1080/17518423.2019.1683907. Epub 2019 Nov 1. PMID 31674852
- [Background] Rathinam C, Mohan V, Peirson J, Skinner J, Nethaji KS, Kuhn I. Effectiveness of virtual reality in the treatment of hand function in children with cerebral palsy: A systematic review. J Hand Ther. 2019 Oct-Dec;32(4):426-434.e1. doi: 10.1016/j.jht.2018.01.006. Epub 2018 Jul 14. PMID 30017414
- [Background] Romero-Ayuso D, Toledano-Gonzalez A, Rodriguez-Martinez MDC, Arroyo-Castillo P, Trivino-Juarez JM, Gonzalez P, Ariza-Vega P, Gonzalez ADP, Segura-Fragoso A. Effectiveness of Virtual Reality-Based Interventions for Children and Adolescents with ADHD: A Systematic Review and Meta-Analysis. Children (Basel). 2021 Jan 21;8(2):70. doi: 10.3390/children8020070. PMID 33494272
- [Background] Burin-Chu S, Baillet H, Leconte P, Lejeune L, Thouvarecq R, Benguigui N. Effectiveness of virtual reality interventions of the upper limb in children and young adults with cerebral palsy: A systematic review with meta-analysis. Clin Rehabil. 2024 Jan;38(1):15-33. doi: 10.1177/02692155231187858. Epub 2023 Jul 27. PMID 37499213
- [Background] Levac DE, Huber ME, Sternad D. Learning and transfer of complex motor skills in virtual reality: a perspective review. J Neuroeng Rehabil. 2019 Oct 18;16(1):121. doi: 10.1186/s12984-019-0587-8. PMID 31627755
- [Background] van den Broek MD. Why does neurorehabilitation fail? J Head Trauma Rehabil. 2005 Sep-Oct;20(5):464-73. doi: 10.1097/00001199-200509000-00007. PMID 16170254
- [Background] Jackman M, Sakzewski L, Morgan C, Boyd RN, Brennan SE, Langdon K, Toovey RAM, Greaves S, Thorley M, Novak I. Interventions to improve physical function for children and young people with cerebral palsy: international clinical practice guideline. Dev Med Child Neurol. 2022 May;64(5):536-549. doi: 10.1111/dmcn.15055. Epub 2021 Sep 21. PMID 34549424
- [Background] Jackman M, Lannin N, Galea C, Sakzewski L, Miller L, Novak I. What is the threshold dose of upper limb training for children with cerebral palsy to improve function? A systematic review. Aust Occup Ther J. 2020 Jun;67(3):269-280. doi: 10.1111/1440-1630.12666. Epub 2020 Apr 27. PMID 32342517
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Wright A, Roberts R, Bowman G, Crettenden A. Barriers and facilitators to physical activity participation for children with physical disability: comparing and contrasting the views of children, young people, and their clinicians. Disabil Rehabil. 2019 Jun;41(13):1499-1507. doi: 10.1080/09638288.2018.1432702. Epub 2018 Jan 30. PMID 29382235
- [Background] Shahmoradi L, Rezayi S. Cognitive rehabilitation in people with autism spectrum disorder: a systematic review of emerging virtual reality-based approaches. J Neuroeng Rehabil. 2022 Aug 18;19(1):91. doi: 10.1186/s12984-022-01069-5. PMID 35982460